CLINICAL TRIAL: NCT06346080
Title: Molecular Analysis for Gastro-Esophageal Cancer: Multicenter Discrete Choice Experiment
Acronym: MAGECmultiDiCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Stijn Vanstraelen, Principal investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: s68670
Record Dates: First submitted 2024-03-23; First posted 2024-04-03 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Esophageal cancer; Survey; Gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A survey will be conducted in a single group of participants from different geographical regions and backgrounds
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey participants (Experimental): Participants who will complete a survey investigating their preference for diagnosis and assessment of gastro-esophageal cancer
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Discrete choice survey

SUMMARY:
The goal of this survey is to investigate the participants' preference for a specific screening/diagnostic tool to detect and assess gastro-esophageal cancer.

The main question it aims to answer are:

* Which diagnostic modality is preferred by patients and the general population?
* Which features of the diagnostic test are most detrimental in the decision-making for one or the other modality?
* Are geographical differences present in regard to the preference for a diagnostic modality?

Participants will be asked to complete a survey of 20-25min, including a brief intake regarding their socio-economic status. This approach will allow us to correct for confounding factors.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals >18yo to 75yo (upper age limit of Barrett's surveillance)
2. Access to computer or smartphone
3. Clear understanding of available languages of the experiment (English, French, Dutch, Spanish, German, Chinese, Japanese)

Exclusion Criteria:

1. Individuals less than 18yo and more than 75yo
2. Incarcerated individuals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of contribution of diagnostic features to the preference of participants | 2 years
  A part-worth analysis, expressed as percentage, from a discrete choice experiment (questionnaire) will assess the features that are most important to the participants
The percentage differences in preference of participants between geographical regions | 2 years
  Differences in preferences will be compared between different geographical regions using chi-squared or McNemar's test

SECONDARY OUTCOMES:
Assess the rate patient-level demographics influence the importance of a test feature, expressed as an odds ratio | 2 years
  Assess the influence of demographic characteristics on the decision-making process using a multivariable logistic regression model, providing odds ratios.
Assess the rate of trade-off demonstrated as odds ratio between cancer-related mortality reduction and costs | 2 years
  Based on an anticipated cancer detection and cost, we will assess the willingness-to-pay using a multivariable logistic regression, providing odds ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Vanstraelen, MD, Principal Investigator — UZ Leuven; Philippe Nafteux, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request with the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code